CLINICAL TRIAL: NCT05264818
Title: Assessment of Endothelial Glycocalyx in Patients With Primary Open-angle Glaucoma: a Prospective Single-center Cross-sectional Case-control Study
Brief Title: Assessment of Endothelial Glycocalyx in Patients With Primary Open-angle Glaucoma
Acronym: GLAUCALYX
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CLL_2021_27
Record Dates: First submitted 2022-02-21; First posted 2022-03-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Primary Open-angle Glaucoma; Glaucoma
Keywords: Glycocheck; Sublingual microvascularization; Glycocalyx; Primary Open-angle Glaucoma; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: primary open angle glaucoma
  Interventions: Procedure: Glycocheck; Procedure: Ophthalmological examinations
- Control group: No Absence of optic nerve pathology
  Interventions: Procedure: Glycocheck; Procedure: Ophthalmological examinations

INTERVENTIONS:
Procedure: Glycocheck — Assessment of the sublingual microvascularization
Procedure: Ophthalmological examinations — Description :
  Measurement of best corrected distance visual acuity with ETDRS (Early Treatment Diabetic Retinopathy Study) Measurement of intraocular pressure by aplanation and forced air tonometer Central corneal thickness measurement with OCT (Optical Coherence Tomography) Non-mydriatic retinophotography Humphrey 24-2 visual field OCT-RNFL (Optical Coherence Tomography - retinal nerve fiber layer)

SUMMARY:
The glycocalyx is a fibrillary lining structure that covers the inner surface of blood vessels. Composed of glycoproteins and polysaccharides, it is an essential determinant of vascular endothelial physiology: it limits coagulation activation and adapts capillary perfusion. Studies have shown glycocalyx alteration in various vascular and autoimmune pathologies such as diabetes, high blood pressure, chronic renal failure, ischemic heart disease, stroke, dementia, septic shock, and several other inflammatory pathologies with a common basis in vascular insufficiency.

Glaucoma is a progressive, chronic and asymptomatic optic neuropathy characterized by visual field damage and abnormalities of the optic nerve head. Two hypotheses have been proposed as a basis for this progressive damage:

* the mechanical theory, which explains the papillary excavation by a compression of the optic nerve head under the effect of high intraocular pressure; and
* the ischemic theory, explained by a circulatory insufficiency at the level of the blood capillaries of the retina and especially of the optic nerve head. This latter theory is related to several pathologies that have circulatory insufficiency as common underlying pathophysiology, and in which damage to the glycocalyx has been well studied.

Glycocalyx damage has rarely been studied in glaucoma. Yang et al. showed that the glycocalyx, present in Schlem's canal, plays a major role in the transduction of shear stress and regulation of outflow resistance to the aqueous humor, which may constitute an interesting biomarker for glaucomatous pathologies.

DETAILED DESCRIPTION:
This study propose to extend the exploration of the ischemic theory of glaucoma by a specific imaging technique (the GlycoCheck) which allows an assessment of the microvascular system integrity by giving a "vitality score" of this system. This score, known as the MicroVascular Health score (MVHS), depends on the following measured parameters: Capillary density (CD), Red blood cell filling Percent (RBF), and Perfused boundary region (PBR).

ELIGIBILITY:
Inclusion Criteria:

* Express consent to participate in the study
* Only for case group: primary open angle glaucoma (defined as the presence of visual field damage attributed to glaucomatous optic neuropathy) in both eyes
* Only for control group: Absence optic nerve pathology (including primary open angle glaucoma)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Sleep apnea
* Renal insufficiency
* Parkinson's disease
* Alzheimer's disease
* Antiphospholipid syndrome
* Cancer for which treatment ended less than 2 years ago
* Stroke less than 1 year ago
* Myocardial infarction less than 1 year ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case group: patients with primary open angle glaucoma Control group : patient with no optic nerve pathology, matched with patients in case group on age (± 10 years), sex (male/female), and smoking status (active smoker/non-smoker or non-smoker or former smoker who had quit smoking for more than 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Thickness of the Perfused boundary region (PBR) | Baseline day
  Evaluated with the Glycocheck, in µm

CONTACTS AND LOCATIONS:
Overall Officials: Cédric LAMIREL, MD, Principal Investigator — Hôpital Fondation A. de Rothschild; Georges AZAR, MD, Study Chair — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France